CLINICAL TRIAL: NCT03894930
Title: Identifying Neural Correlates of Altruism
Brief Title: Metta Meditation Training on Prosocial Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-180; BCS-1729406 (Other Grant/Funding Number: NSF)
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-07

CONDITIONS: Social Behavior
Keywords: healthy subjects; prosocial; metta meditation; fMRI
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metta meditation (Experimental): Eight-week, guided metta meditation training that is administered online
  Interventions: Behavioral: Metta meditation
- Wait-list (No Intervention): Eight-week wait-list control with no training

INTERVENTIONS:
Behavioral: Metta meditation — Administered 5 days per week for 8 weeks.
  Other Names: Loving-kindness meditation
  Arms: Metta meditation

SUMMARY:
The purpose of the study is to look at the impact of a metta meditation training on prosocial behavior and socio-affective brain responses. The training involves an 8-week, online administration of guided metta meditation practices aimed at generating feelings of kindness and compassion for other people. The study examines how participants respond to thinking about familiar others and strangers using behavioral and brain-imaging measures. This study will be important for understanding how people develop the capacity to be prosocial towards other individuals, which is a key component of adaptive social behavior.

ELIGIBILITY:
Inclusion Criteria:

* Is a medically healthy individual
* Lives in the Washington, D.C. metro area and is able to travel to Georgetown University

Exclusion Criteria:

* Has experience with meditation
* Has any MRI contraindication (e.g. metal in the body, cardiac pacemaker, cannot lie still, etc.)
* Has any neurological disease
* Has a current psychiatric disorder
* Is pregnant or planning to become pregnant
* Is on medication that affects the central nervous system (e.g. psychotropic drugs)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Social Discounting | 8 weeks
  During functional magnetic resonance imaging (fMRI) scanning, participants will complete a social discounting task. Participants will choose whether to forgo various amounts of money to give to another person. Behavioral and brain responses will be analyzed to assess social discounting in each participant.
Affective Brain Responses to Familiar and Unfamiliar Others | 8 weeks
  During functional magnetic resonance imaging (fMRI) scanning, participants will view images of people who they know and people who they do not know. Affective brain response patterns will be analyzed to assess responding in each participant.

SECONDARY OUTCOMES:
State Affect Rating | 8 weeks
  Participants will complete the Positive Affect Negative Affect Schedule (PANAS) questionnaire. This self-report scale includes 20 items that are rated on a 5-point scale of 1 (not at all) to 5 (very much). Positive and negative self-reported affect will be quantified for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail A Marsh, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No